CLINICAL TRIAL: NCT02006472
Title: A Phase 2, Dose-Finding, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled Study, Evaluating the Safety and Efficacy of Pridopidine 45, 67.5, 90, and 112.5 mg Twice-Daily vs Placebo for Symptomatic Treatment in Patients With Huntington's Disease
Brief Title: A Phase 2, to Evaluating the Safety and Efficacy of Pridopidine Vs Placebo for Symptomatic Treatment in Patients With Huntington's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prilenia (Industry)
Collaborators: European Huntington's Disease Network (Network); Huntington Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV7820-CNS-20002; 2013-001888-23 (EudraCT Number)
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-05

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease; Pridopidine; Pride-HD
MeSH Terms: conditions — Huntington Disease | interventions — pridopidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Pridopidine 45 mg (Experimental): Twice daily
  Interventions: Drug: Pridopidine; Other: Placebo
- Pridopidine 67.5 mg (Experimental): Twice daily
  Interventions: Drug: Pridopidine; Other: Placebo
- Pridopidine 90 mg (Experimental): Twice daily
  Interventions: Drug: Pridopidine; Other: Placebo
- Pridopidine 112.5 mg (Experimental): Twice daily
  Interventions: Drug: Pridopidine; Other: Placebo
- Placebo (Placebo Comparator): Twice daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pridopidine — 22.5 mg and 45 mg capsules
  Other Names: TV7820
  Arms: Pridopidine 112.5 mg; Pridopidine 45 mg; Pridopidine 67.5 mg; Pridopidine 90 mg
Other: Placebo — Capsules matching drug

SUMMARY:
This is a multicenter, multinational, randomized, parallel-group, double-blind, placebo-controlled, dose range finding study to compare the efficacy and safety of different doses of pridopidine versus placebo in the treatment of motor impairment in Huntington's Disease (HD).

DETAILED DESCRIPTION:
Originally, the study was designed to assess the effect of pridopidine on motor function at 26 weeks. Due to the recognition that the primary target of pridopidine is the Sigma-1 receptor, the trial was extended from 26 to 52 weeks to evaluate the effect of pridopidine on Total Functional Capacity (TFC). A minimum of 52 weeks are needed for the placebo group to decline and allow a window to assess an effect on TFC (a prespecified endpoint). Approximately 20% of patients completed 26 weeks of the study before IRB approvals for this extension, and did not continue into the 2nd treatment period up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HD based on the presence of >/= 36 CAG repeats
* Male or female age ≥21 years, with an onset of HD after 18 years' old.
* Females of childbearing potential must be compliant in using adequate birth control throughout the duration of the study
* Body weight ≥50 kg
* Sum of >= 25 points on the UHDRS-TMS and UHDRS Independence Score <=90%
* Able and willing to provide written informed consent prior to any study related procedure.
* Willing to provide a blood sample for genetic analyses
* Willing and able to take oral medication and able to comply with the study specific procedures.
* Ambulatory, being able to travel to the study center, and judged by the investigator as likely to be able to continue to travel for the duration of the study.
* Availability and willingness of a caregiver, informant or family member to accompany the patient to the clinic at study, and the suitability of the caregiver should be judged by the Investigator.

  * Other criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* Patients with clinically significant heart disease at the screening visit
* Treatment with tetrabenazine within 6 weeks of study screening
* Patients with a history of epilepsy or of seizures within the last 5 years
* Have other serious medical illnesses in the opinion of the investigator may put the patient at risk when participating in the study or may influence the results of the study or affect the patient's ability to take part in the study
* Patients receiving medications (within the last 6 weeks prior to screening) that have been proven to prolong QT interval or who may require such medications during the course of the study such as but not limited to non allowed anti psychotic medications, tricyclic antidepressants and/or Class I antiarrhythmics

  * Other criteria apply, please contact the investigator for more information

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2015-12-16 (Actual); Study Completion 2016-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (58):
- United States (16):
  - Investigational Site 12199, La Jolla, California
  - Investigational Site 12204, Los Angeles, California
  - Investigational Site 12201, Englewood, Colorado
  - Investigational Site 12196, Washington D.C., District of Columbia
  - Investigational Site 12207, Chicago, Illinois
  - Investigational Site 12202, Baltimore, Maryland
  - Investigational Site 12206, Baltimore, Maryland
  - Investigational Site 12200, Manhasset, New York
  - Investigational Site 12203, New York, New York
  - Investigational Site 12198, Rochester, New York
  - Investigational Site 12211, Winston-Salem, North Carolina
  - Investigational Site 12205, Cincinnati, Ohio
  - Investigational Site 12209, Pittsburgh, Pennsylvania
  - Investigational Site 12208, Salt Lake City, Utah
  - Investigational Site 12210, Richmond, Virginia
  - Investigational Site 12197, Kirkland, Washington
- Australia (4):
  - Investigational Site 78055, Caulfield South
  - Investigational Site 78056, Kew
  - Investigational Site 78058, Subiaco
  - Investigational Site 78057, Westmead
- Austria (2):
  - Investigational Site 33021, Innsbruck
  - Investigational Site 33027, Vienna
- Canada (3):
  - Investigational Site 11035, Vancouver, British Columbia
  - Investigational Site 11037, Ottawa, Ontario
  - Investigational Site 11036, Toronto, Ontario
- Denmark (2):
  - Investigational Site 39028, Aarhus
  - Investigational Site 39027, Copenhagen
- France (6):
  - Investigational Site 35123, Angers
  - Investigational Site 35122, Créteil
  - Investigational Site 35125, Lille
  - Investigational Site 35124, Marseille
  - Investigational Site 35121, Salouël
  - Investigational Site 35165, Toulouse
- Germany (4):
  - Investigational Site 32408, Berlin
  - Investigational Site 32410, Bochum
  - Investigational Site 32409, Münster
  - Investigational Site 32407, Ulm
- Italy (5):
  - Investigational Site 30083, Florence
  - Investigational Site 30080, Milan
  - Investigational Site 30082, Napoli
  - Investigational Site 30081, Pozzilli
  - Investigational Site 30084, San Giovanni Rotondo
- Investigational Site 38059, Leiden, Netherlands
- Poland (4):
  - Investigational Site 53150, Gdansk
  - Investigational Site 53149, Krakow
  - Investigational Site 53148, Poznan
  - Investigational Site 53151, Warsaw
- Russia (3):
  - Investigational Site 50215, Kazan'
  - Investigational Site 50213, Moscow
  - Investigational Site 50214, Nizhny Novgorod
- United Kingdom (8):
  - Investigational Site 34058, Birmingham
  - Investigational Site 34054, Cambridge
  - Investigational Site 34059, Cardiff
  - Investigational Site 34056, Headington
  - Investigational Site 34060, London
  - Investigational Site 34055, Manchester
  - Investigational Site 34061, Newcastle upon Tyne
  - Investigational Site 34057, Sheffield

REFERENCES:
- [Background] McGarry A, Leinonen M, Kieburtz K, Geva M, Olanow CW, Hayden M. Effects of Pridopidine on Functional Capacity in Early-Stage Participants from the PRIDE-HD Study. J Huntingtons Dis. 2020;9(4):371-380. doi: 10.3233/JHD-200440. PMID 33164941
- [Derived] Darpo B, Geva M, Ferber G, Goldberg YP, Cruz-Herranz A, Mehra M, Kovacs R, Hayden MR. Pridopidine Does Not Significantly Prolong the QTc Interval at the Clinically Relevant Therapeutic Dose. Neurol Ther. 2023 Apr;12(2):597-617. doi: 10.1007/s40120-023-00449-w. Epub 2023 Feb 22. PMID 36811812
- [Derived] Rodrigues FB, Quinn L, Wild EJ. Huntington's Disease Clinical Trials Corner: January 2019. J Huntingtons Dis. 2019;8(1):115-125. doi: 10.3233/JHD-190001. PMID 30776019
- [Derived] Reilmann R, McGarry A, Grachev ID, Savola JM, Borowsky B, Eyal E, Gross N, Langbehn D, Schubert R, Wickenberg AT, Papapetropoulos S, Hayden M, Squitieri F, Kieburtz K, Landwehrmeyer GB; European Huntington's Disease Network; Huntington Study Group investigators. Safety and efficacy of pridopidine in patients with Huntington's disease (PRIDE-HD): a phase 2, randomised, placebo-controlled, multicentre, dose-ranging study. Lancet Neurol. 2019 Feb;18(2):165-176. doi: 10.1016/S1474-4422(18)30391-0. Epub 2018 Dec 15. PMID 30563778

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 492 patients were screened; of these, 408 were randomized. The main reason for not randomizing patients was noncompliance with the eligibility criteria.
Groups:
- Placebo: Pridopidine matching placebo (hard capsules)
  Patients received a starting dose of placebo matching pridopidine 22.5 mg and were during the first 4 weeks of treatment titrated to the randomized dose level. The randomized dose level was then to be maintained for the remainder of the treatment period through Week 52.
- Pridopidine 45 mg BID; Pridopidine 67.5 mg BID; Pridopidine 90 mg BID; Pridopidine 112.5 mg BID: Pridopidine given as hard capsules, twice daily
  Patients received a starting dose of pridopidine 22.5 mg and were during the first 4 weeks of treatment titrated to their randomized dose level. The randomized dose level was then to be maintained for the remainder of the treatment period through Week 52.
Period: Period 1 (Through Week 26)
Arm/Group | Placebo | Pridopidine 45 mg BID | Pridopidine 67.5 mg BID | Pridopidine 90 mg BID | Pridopidine 112.5 mg BID
Started | 82 | 81 | 82 | 81 | 82
ITT (Intention-to-treat: patients randomised into the study and dispensed study drug.) | 82 | 81 | 82 | 81 | 82
FAS (Full analysis set: patients from the ITT who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment. The FAS included efficacy observations measured up to Week 52.) | 81 | 75 | 79 | 81 | 81
Safety Set (Including all patients who took at least 1 dose of study drug. The analysis set included safety observations measured up to Week 52.) | 82 | 81 | 82 | 81 | 82
Completed | 70 | 59 | 65 | 67 | 62
Not Completed | 12 | 22 | 17 | 14 | 20
Not completed — Protocol Violation | 1 | 1 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0
Not completed — Noncompliance | 2 | 1 | 1 | 0 | 0
Not completed — Other | 1 | 5 | 0 | 2 | 3
Not completed — Adverse Event | 5 | 6 | 11 | 11 | 14
Not completed — Withdrawal by Subject | 3 | 9 | 3 | 0 | 3
Period: Period 2 (Through Week 52)
Arm/Group | Placebo | Pridopidine 45 mg BID | Pridopidine 67.5 mg BID | Pridopidine 90 mg BID | Pridopidine 112.5 mg BID
Started (The trial was extended from 26 to 52 weeks to evaluate the effect of pridopidine on Total Functional Capacity (TFC). Approximately 20% of patients completed 26 weeks of the study before IRB approvals for this extension, and did not continue into the 2nd treatment period up to 52 weeks.) | 57 | 49 | 54 | 56 | 46
Started Treatment in Period 2 | 57 | 49 | 52 | 56 | 46
Completed | 52 | 43 | 44 | 53 | 44
Not Completed | 5 | 6 | 10 | 3 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1 | 1
Not completed — Noncompliance | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 4 | 5 | 1 | 1
Not completed — Other | 0 | 1 | 0 | 1 | 0
Not completed — Not treated | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 0 | 0
Not completed — Sponsor decision | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat: all patients randomized into the study
Groups:
- Placebo: Pridopidine matching placebo (hard capsules)
  Patients received a starting dose of placebo matching pridopidine 22.5 mg or matching placebo and were during the first 4 weeks of treatment titrated to their randomized dose level. The randomized dose level was then to be maintained for the remainder of the treatment period through Week 52.
- Total: Total of all reporting groups
Arm/Group | Placebo | Pridopidine 45 mg BID | Pridopidine 67.5 mg BID | Pridopidine 90 mg BID | Pridopidine 112.5 mg BID | Total
Number analyzed (Participants) | 82 | 81 | 82 | 81 | 82 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (11.34) | 51.9 (11.75) | 51.0 (11.83) | 51.3 (12.69) | 47.5 (11.40) | 50.4 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 41 | 43 | 39 | 203
  Male | 42 | 41 | 41 | 38 | 43 | 205
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 73 | 75 | 78 | 75 | 77 | 378
  Black | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1 | 0 | 2
  Other | 0 | 1 | 0 | 1 | 0 | 2
  Missing | 8 | 5 | 3 | 4 | 5 | 25
Use of neuroleptics [Count of Participants; unit: Participants]
  Yes | 31 | 31 | 32 | 31 | 32 | 157
  No | 51 | 50 | 50 | 50 | 50 | 251
CYP2D6 genotype [Count of Participants; unit: Participants]
  Poor metaboliser | 1 | 5 | 4 | 2 | 4 | 16
  Extensive metaboliser | 72 | 70 | 70 | 74 | 69 | 355
  Intermediate metaboliser | 8 | 5 | 8 | 5 | 9 | 35
  Ultra-rapid metaboliser | 1 | 1 | 0 | 0 | 0 | 2
Number of Cytosine-Adenosine-Guanine (CAG) Repeats [Mean (Standard Deviation); unit: Number of CAG repeats] | 44.4 (3.23) | 44.1 (4.12) | 45.0 (4.73) | 44.5 (4.90) | 45.3 (3.66) | 44.7 (4.18)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale-Total Motor Score (UHDRS-TMS) at Week 26
Description: TMS was defined as the sum of all UHDRS motor domains ratings. The motor section of the UHDRS assesses motor features of Huntington's Disease (HD) with standardized ratings of oculo-motor function, dysarthria, chorea, dystonia, gait, and postural stability. Each of 15 assessments is rated on a scale of 0 (normal) to 4 (marked impairment) for a TMS range of 0-124. Negative change from baseline values indicate improvement.
Time Frame: 26 weeks
Population: Full analysis set (FAS) i.e. patients who received at least one dose of study drug and had at least one post-baseline efficacy assessment
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Pridopidine matching placebo (hard capsules)
  Patients received a starting dose of placebo matching pridopidine 22.5 mg and were during the first 4 weeks of treatment titrated to their randomized dose level. The randomized dose level was then to be maintained for the remainder of the treatment period through Week 52.
Arm/Group | Placebo | Pridopidine 45 mg BID | Pridopidine 67.5 mg BID | Pridopidine 90 mg BID | Pridopidine 112.5 mg BID
Number analyzed (Participants) | 81 | 75 | 79 | 81 | 81
score on a scale | -4.79 (0.99) | -3.37 (1.05) | -3.09 (1.02) | -4.13 (1.00) | -2.74 (1.01)
Statistical Analysis 1: Comparison: Placebo vs Pridopidine 45 mg BID; Test type: Superiority; p = 0.3202, Mixed Models Analysis; LSM difference = 1.42, 95% CI 2-sided [-1.39 to 4.23]
Statistical Analysis 2: Comparison: Placebo vs Pridopidine 67.5 mg BID; Test type: Superiority; p = 0.2266, Mixed Models Analysis; LSM difference = 1.7, 95% CI 2-sided [-1.06 to 4.46]
Statistical Analysis 3: Comparison: Placebo vs Pridopidine 90 mg BID; Test type: Superiority; p = 0.6348, Mixed Models Analysis; LSM difference = 0.66, 95% CI 2-sided [-2.07 to 3.39]
Statistical Analysis 4: Comparison: Placebo vs Pridopidine 112.5 mg BID; Test type: Superiority; p = 0.1447, Mixed Models Analysis; LSM difference = 2.04, 95% CI 2-sided [-0.71 to 4.8]

2. Secondary Outcome: Number of Patients With Adverse Events
Time Frame: 52 weeks
Population: Safety Analysis set, i.e. patients who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Pridopidine matching placebo (hard capsules)
  Patients received a starting dose of pridopidine 22.5 mg or matching placebo and were during the first 4 weeks of treatment titrated to their randomised dose level. The randomised dose level was then to be maintained for the remainder of the treatment period through Week 52.
- Pridopidine 45 mg BID; Pridopidine 67.5 mg BID; Pridopidine 90 mg BID; Pridopidine 112.5 mg BID: Pridopidine given as hard capsules, twice daily
  Patients received a starting dose of pridopidine 22.5 mg (or matching placebo) and were during the first 4 weeks of treatment titrated to their randomised dose level. The randomised dose level was then to be maintained for the remainder of the treatment period through Week 52.
Arm/Group | Placebo | Pridopidine 45 mg BID | Pridopidine 67.5 mg BID | Pridopidine 90 mg BID | Pridopidine 112.5 mg BID
Number analyzed (Participants) | 82 | 81 | 82 | 81 | 82
Participants | 62 | 63 | 69 | 71 | 67

3. Other Pre Specified Outcome: Change From Baseline in Total Functional Capacity (TFC) at Week 52
Description: The TFC is one subscale of the Unified Huntington's Disease Rating Scale (UHDRS), comprising 5 functional domains associated with disability (occupation, finances, domestic chores, activities of daily living, and care level), with scores on each item ranging from 0 to either 2 or 3. The TFC total score is the sum of the 5 TFC items and can range from 0 to 13, with greater scores indicating higher functioning. Negative change from baseline indicates worsening.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Pridopidine 45 mg BID | Pridopidine 67.5 mg BID | Pridopidine 90 mg BID | Pridopidine 112.5 mg BID
Number analyzed (Participants) | 81 | 75 | 78 | 81 | 81
score on a scale | -0.83 (0.20) | 0.04 (0.22) | -0.72 (0.21) | -0.65 (0.20) | -0.59 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Pridopidine 45 mg BID; Test type: Superiority; p = 0.0032, Mixed Models Analysis; LSM difference = 0.87, 95% CI 2-sided [0.29 to 1.45]
Statistical Analysis 2: Comparison: Placebo vs Pridopidine 67.5 mg BID; Test type: Superiority; p = 0.7042, Mixed Models Analysis; LSM difference = 0.11, 95% CI 2-sided [-0.46 to 0.68]
Statistical Analysis 3: Comparison: Placebo vs Pridopidine 90 mg BID; Test type: Superiority; p = 0.5099, Mixed Models Analysis; LSM difference = 0.19, 95% CI 2-sided [-0.37 to 0.75]
Statistical Analysis 4: Comparison: Placebo vs Pridopidine 112.5 mg BID; Test type: Superiority; p = 0.4061, Mixed Models Analysis; LSM difference = 0.24, 95% CI 2-sided [-0.33 to 0.82]

4. Post Hoc Outcome: Change in Total Functional Capacity (TFC) From Baseline in Patients With Early HD (Defined as Patients With TFC>=7)
Description: as for outcome 3
Time Frame: 52 weeks
Population: FAS i.e. pts receiving ≥1 dose of study drug and with ≥1 post-BL efficacy assessment; pts with early HD defined by BL TFC score ≥7.
  The study tested 4 pridopidine doses on TMS for 26 w. Due to a new understanding on pridopidine's mechanism of action (S1R agonist), the study was extended to 52w to assess TFC in all HD. A post-hoc analysis for the 45 mg bid dose was performed for TFC in early HD, and the dose was chosen for Phase 3.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Pridopidine 45 mg BID
Number analyzed (Participants) | 62 | 59
score on a scale | -1.17 (0.22) | -0.01 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Pridopidine 45 mg BID; Test type: Superiority; p = 0.0003, Mixed Models Analysis; LSM difference = 1.16, 95% CI 2-sided [0.54 to 1.78]

5. Post Hoc Outcome: Total Functional Capacity Responder Rate in Early HD
Description: The TFC is one subscale of the Unified Huntington's Disease Rating Scale (UHDRS), comprising 5 functional domains associated with disability (occupation, finances, domestic chores, activities of daily living, and care level), with scores on each item ranging from 0 to either 2 or 3. The TFC total score is the sum of the 5 TFC items and can range from 0 to 13, with greater scores indicating higher functioning.
  Responder was defined as a TFC change to Week 52 of TFC>=0.
Time Frame: 52 weeks
Population: FAS i.e. pts receiving ≥1 dose of study drug and with ≥1 post-BL efficacy assessment; pts with early HD defined by BL TFC score ≥7 who completed 52 weeks.
  The study tested 4 pridopidine doses on TMS for 26 w. Due to a new understanding on pridopidine's mechanism of action (S1R agonist), the study was extended to 52w to assess TFC in all HD. A post-hoc analysis for the 45 mg bid dose was performed for TFC in early HD, and the dose was chosen for Phase 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pridopidine 45 mg BID
Number analyzed (Participants) | 41 | 37
Participants | 20 | 30
Statistical Analysis 1: Comparison: Placebo vs Pridopidine 45 mg BID; Test type: Superiority; p = 0.003, Chi-squared

6. Post Hoc Outcome: Change From Baseline in Quantitative Motor (Q-motor) Measurements, Pro-Sup-Inter-Tap-interval-MN-Hand, Early HD
Description: Q-motor assessments were based on the application of force transducers and 3-dimensional position sensors. The reported parameter is the Pro-Sup-Inter-Tap-interval-MN-Hand, measured in seconds. Positive change from baseline indicates worsening.
Time Frame: 26 and 52 weeks
Population: FAS i.e. pts receiving >=1 dose of study drug and with >=1 post-BL efficacy assessment; pts with early HD defined by BL TFC score ≥7.
  The study tested 4 pridopidine doses on TMS for 26 w. Due to a new understanding on pridopidine's mechanism of action (S1R agonist), the study was extended to 52w to assess TFC in all HD. A post-hoc analysis for the 45 mg bid dose was performed for TFC in early HD, and the dose was chosen for Phase 3.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Pridopidine 45 mg BID
Number analyzed (Participants) | 62 | 59
seconds
  Change from baseline to Week 26 | 0.0247 (0.0118) | -0.0096 (0.0110)
  Change from baseline to Week 52 | 0.0447 (0.0142) | 0.0003 (0.0150)
Statistical Analysis 1: Comparison: Placebo vs Pridopidine 45 mg BID; At Week 26; Test type: Superiority; p = 0.0346, Mixed Models Analysis; LSM difference = -0.0341, 95% CI 2-sided [-0.0658 to -0.0026]
Statistical Analysis 2: Comparison: Placebo vs Pridopidine 45 mg BID; At Week 52; Test type: Superiority; p = 0.0305, Mixed Models Analysis; LSM difference = -0.0444, 95% CI 2-sided [-0.0847 to -0.0042]

ADVERSE EVENTS:
Time Frame: 52 weeks
Groups:
- Placebo: Pridopidine matching placebo (hard capsules)
  Patients received a starting dose of pridopidine 22.5 mg or matching placebo and were during the first 4 weeks of treatment titrated to their randomised dose level. The randomised dose level was then to be maintained for the remainder of the treatment period through Week 26.
- Pridopidine 45 mg BID; Pridopidine 67.5 mg BID; Pridopidine 90 mg BID; Pridopidine 112.5 mg BID: Pridopidine given as hard capsules, twice daily
  Patients received a starting dose of pridopidine 22.5 mg (or matching placebo) and were during the first 4 weeks of treatment titrated to their randomised dose level. The randomised dose level was then to be maintained for the remainder of the treatment period through Week 26.
Arm/Group | Placebo | Pridopidine 45 mg BID | Pridopidine 67.5 mg BID | Pridopidine 90 mg BID | Pridopidine 112.5 mg BID
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/81 | 0/82 | 1/81 | 1/82
Serious Adverse Events (participants affected / at risk) | 0/82 | 8/81 | 9/82 | 9/81 | 9/82
Other Adverse Events (participants affected / at risk) | 45/82 | 49/81 | 63/82 | 57/81 | 53/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Pridopidine 45 mg BID (N=81) | Pridopidine 67.5 mg BID (N=82) | Pridopidine 90 mg BID (N=81) | Pridopidine 112.5 mg BID (N=82)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of the colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tetention (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Pridopidine 45 mg BID (N=81) | Pridopidine 67.5 mg BID (N=82) | Pridopidine 90 mg BID (N=81) | Pridopidine 112.5 mg BID (N=82)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (6) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 17 (31) | 16 (44) | 21 (31) | 13 (19) | 16 (42)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 6 (7) | 6 (8) | 0 (0) | 3 (4)
Weight decreased (Investigations) | 3 (3) | 4 (4) | 3 (3) | 3 (3) | 7 (7)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 5 (6) | 2 (2) | 3 (4) | 5 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 2 (2) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 8 (8) | 7 (18) | 7 (11) | 11 (19) | 8 (10)
Chorea (Nervous system disorders) | 1 (1) | 4 (4) | 13 (15) | 3 (3) | 7 (8)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 6 (12) | 5 (5) | 6 (8)
Balance disorder (Nervous system disorders) | 3 (3) | 2 (3) | 5 (6) | 1 (1) | 3 (3)
Fatigue (General disorders) | 7 (10) | 3 (3) | 6 (6) | 7 (8) | 5 (5)
Anxiety (Psychiatric disorders) | 2 (2) | 6 (6) | 6 (6) | 7 (8) | 5 (5)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 7 (8) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (5) | 5 (6) | 11 (11) | 9 (10) | 9 (11)
Irritability (Psychiatric disorders) | 7 (8) | 4 (4) | 6 (7) | 5 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (14) | 9 (11) | 11 (14) | 11 (17) | 10 (15)
Vomiting (Gastrointestinal disorders) | 4 (6) | 5 (7) | 6 (7) | 5 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (6) | 7 (10) | 4 (6) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 3 (3) | 6 (9) | 5 (6)
Nasopharyngitis (Infections and infestations) | 7 (8) | 14 (21) | 12 (16) | 13 (15) | 15 (23)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3) | 6 (6) | 4 (5) | 5 (6)

LIMITATIONS AND CAVEATS:
Analyses for Early HD population were conducted as additional analyses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data and results are owned by the sponsor. Results can be used by the institution for (a) internal noncommercial research, education and patient care, and (b) as required under applicable laws and regulations. Other uses require prior written consent of the sponsor.